CLINICAL TRIAL: NCT06821698
Title: An Open-label Study to Determine the Effect of Oral Doses of KP-001 on Rosuvastatin and Caffeine PK After a Single Oral Administration and to Determine the Effect of Fluvoxamine on KP-001 PK After a Single Oral Administration in Volunteers
Brief Title: To Determine the Effect of KP-001 on Rosuvastatin, Caffeine PK and the Effect of Fluvoxamine on KP-001 PK in Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kaken Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KP-001-106
Record Dates: First submitted 2025-02-06; First posted 2025-02-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Healty Volunteers
MeSH Terms: interventions — caffeine citrate; Fluvoxamine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- KP-001/Rosuvastatin calcium (Experimental)
  Interventions: Drug: KP-001; Drug: Rosuvastatin calcium10mg
- KP-001/Caffeine citrate (Experimental)
  Interventions: Drug: KP-001; Drug: Caffeine citrate
- KP-001/Fluvoxamine (Experimental)
  Interventions: Drug: KP-001; Drug: Fluvoxamine

INTERVENTIONS:
Drug: KP-001 — KP-001 100 mg dry syrup
Drug: Rosuvastatin calcium10mg — A oral dose of 10 mg tablet
  Arms: KP-001/Rosuvastatin calcium
Drug: Caffeine citrate — 100 mg oral solution
  Arms: KP-001/Caffeine citrate
Drug: Fluvoxamine — 50 mg tablet
  Arms: KP-001/Fluvoxamine

SUMMARY:
Part 1 will evaluate the effects of KP-001 as an inhibitor of BCRP on the PK of rosuvastatin. In the Treatment Period 1, a single dose of rosuvastatin will be administered. In the Treatment Period 2, KP-001 will be administered once daily for 7 days and a single dose of rosuvastatin will be administered. Blood PK assessments of rosuvastatin will be performed until 48 hours postdose in each Treatment Period. Part 2 will evaluate the effects of KP-001 as an inducer and inhibitor of CYP1A2 on the PK of caffeine. A single dose of caffeine will be administered in the Treatment Period 1. KP-001 will be administered once daily for 10 days and a single dose of caffeine will be administered in the Treatment Period 2. Blood PK assessments of caffeine will be performed until 24 hours postdose in each Treatment Period. Part 3 will evaluate the effects of fluvoxamine as an inhibitor of CYP1A2 on the PK of KP-001. A single dose of KP-001 will be administered in the Treatment Period 1. Fluvoxamine will be administered as a single dose on the first day and then twice daily for 5 days and a single dose of KP-001 will be administered in the Treatment Period 2. Blood PK assessments of KP-001 will be performed until 48 hours postdose in each Treatment Period.

ELIGIBILITY:
Inclusion Criteria:

1. A participant who voluntarily agrees to participate in this study and signs an IRB-approved informed consent prior to performing any of the Screening Visit procedures.
2. A male or female participant who is between 18 to 55 years of age, inclusive, at the Screening Visit.
3. (Part 1 only) A participant who is non-Asian.
4. A female participant who is non-childbearing potential defined in Section 10.4 and not pregnant or breastfeeding.
5. A male participant who is sexually active with female partner(s) of childbearing potential must agree to use both a condom and spermicide from the first dose until 91 days after the last dose of KP-001.
6. A male participant who agrees not to donate sperm from the first dose until 91 days after the last dose of KP-001.
7. A continuous nonsmoker who has not used nicotine-containing products for at least 3 months prior to Day -1 of Treatment Period 1 and throughout the study, based on participant self-reporting and the result of cotinine test at screening and/or Day -1 of each Treatment Period.
8. A participant who is medically healthy with no clinically significant abnormal screening results (eg, medical history, physical examination, laboratory profiles, vital signs, or ECGs), in the opinion of the Investigator or designee. If screening and/or admission results are abnormal, they may be repeated once at screening and/or once at admission to confirm the participant's eligibility.
9. A participant who has body weight ≥ 50.0 kg and body mass index within the range 18.0 to 30.0 kg/m2, inclusive, at the Screening Visit.

Exclusion Criteria:

1. A participant who is legally, mentally or physically incapacitated or, in the opinion of the Investigator, has significant mental or emotional problems, including psychiatric illness (eg, depression and/or anxiety) at the time of the Screening Visit, or that could reasonably be expected to develop during the conduct of the study.
2. A participant with significant history or clinical manifestation of any metabolic, allergic, dermatologic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder as determined by the Investigator or designee.
3. A participant with a history of any illness that, in the opinion of the Investigator or designee, might confound the results of the study or poses an additional risk to the participant by their participation in the study.
4. (For Part 3 only) A participant who meets any of the following criteria based on the C-SSRS assessment at screening:

   1. Presence of suicidal ideation within the 6 months prior to screening (an answer of "yes" on Questions 1 or 2 of the C-SSRS Baseline/Screening version)
   2. Any lifetime history of suicidal ideation (an answer of "yes" on Questions 4 or 5 of the C-SSRS Baseline/Screening version).
   3. Any lifetime history of suicidal behavior as detected by the C-SSRS Baseline/Screening version.
5. A participant who used any prescription or non-prescription medications (including vitamins, recreational drugs, and dietary or herbal supplements) within 14 days or 5 half-lives (whichever is longer) prior to Day -1 of Treatment Period 1 and until completion of the Follow-up Call unless, in the opinion of the Investigator, may be treatment for an AE or will not interfere with the interpretation of safety or the PK assessments.
6. A participant who underwent blood donation or transfusion within 56 days prior to Day -1 of Treatment Period 1 and throughout the study.
7. A participant with a history or presence of hypersensitivity or idiosyncratic reaction to any components of the KP-001 formulation or any components of formulation used as study intervention during the study.
8. A participant with a history of drug or alcohol abuse (regular alcohol consumption exceeding 14 drinks/week [1 drink=5 ounces of wine, 12 ounces of beer, or 1.5 ounces of hard liquor]) within one year before the Screening Visit.
9. A participant who has enrolled in any clinical study of KP-001.
10. A participant with a complication of drug allergies or a history of drug allergies.
11. A participant who used any investigational drug in the last 30 days or 5 half-lives (if known), whichever is longer, prior to Day -1 of Treatment Period 1.
12. A participant who had any major illness within 30 days before the Screening Visit.
13. A participant who had any major surgical procedure within 30 days prior to Day -1 of Treatment Period 1 or any planned surgery during the study period.
14. A participant who had any laboratory abnormality that, in the judgment of the Investigator, would put the participant at unacceptable risk for participation in the study or may interfere with the assessments included in the study.
15. A participant with abnormal findings on the screening ECG deemed clinically significant by the Investigator or qualified designee.
16. A participant who is an employee of the Sponsor or any CRO involved in the study, the Investigator, or an immediate family member (partner, offspring, parents, siblings, or sibling's offspring) of an employee involved in the study.
17. (Part 2) A participant who has consumed alcohol- or caffeine-containing foods and beverages (eg, coffee, tea, cola, soda, cocoa, chocolate, and energy drink) within 72 hours prior to Day -1 of Treatment Period 1 and does not agree to refrain from consuming during the entire study. (Parts 1 and 3) A participant who has consumed alcohol- or caffeine-containing foods and beverages (eg, coffee, tea, cola, soda, cocoa, chocolate, and energy drink) within 72 hours prior to Day -1 of Treatment Period 1 and does not agree to refrain from consuming during the entire study, unless deemed acceptable by the Investigator.
18. A participant with positive urine drug or urine alcohol and positive cotinine test results at screening or Day -1 of Treatment Period 1.
19. A participant who has consumed grapefruit-containing foods and beverages within 7 days prior to Day -1 of Treatment Period 1 and does not agree to refrain from consuming during the entire study.
20. A participant who has consumed St. John's wort-containing foods and beverages within 14 days prior to Day -1 of Treatment Period 1 and does not agree to refrain from consuming during the entire study.
21. A participant who is unable or unwilling to undergo multiple venipunctures.
22. A participant with a history or presence of liver disease or cholecystectomy within one year prior to screening.
23. A participant with an HbA1c >5.7% at screening.
24. A participant with positive results at screening for human immunodeficiency virus, hepatitis B core antibody, hepatitis B surface antigen or hepatitis C virus.
25. A participant with a disorder or any condition that would interfere with the absorption, distribution, metabolism, or excretion of drugs.
26. A participant with an eGFR calculated using the CKD-EPI formula <80 mL/min at screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2025-02-13 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
PK parameters of rosuvastatin in plasma: AUCinf | 48hour
PK parameters of rosuvastatin in plasma: Cmax | 48hour
PK parameters of caffeine in plasma: AUCinf | 24hour
PK parameters of caffeine in plasma: Cmax | 24hour
PK parameters of KP-001 in plasma: AUCinf | 48hour
PK parameters of KP-001 in plasma: Cmax | 48hour

SECONDARY OUTCOMES:
PK parameters of rosuvastatin in plasma: AUClast | 48hour
PK parameters of rosuvastatin in plasma: Tmax | 48hour
PK parameters of rosuvastatin in plasma: t1/2 | 48hour
PK parameters of rosuvastatin in plasma: CLtot/F | 48hour
PK parameters of rosuvastatin in plasma: Vz/F | 48hour
PK parameters of caffeine in plasma: AUClast | 24hour
PK parameters of caffeine in plasma: t1/2 | 24hour
PK parameters of caffeine in plasma: Tmax | 24hour
PK parameters of caffeine in plasma: CLtot/F | 24hour
PK parameters of caffeine in plasma: Vz/F | 24hour
PK parameters of KP-001 in plasma: AUClast | 48hour
PK parameters of KP-001 in plasma: Tmax | 48hour
PK parameters of KP-001 in plasma: t1/2 | 48hour
PK parameters of KP-001 in plasma: Vz/F | 48hour

CONTACTS AND LOCATIONS:
Locations (1):
- Parexel International Early Phase Clinical Unit, Glendale, California, United States